CLINICAL TRIAL: NCT03875469
Title: Performance of Centargo - A Novel Piston-based Injection System for High Throughput in Contrast-enhanced Computed Tomography (CE CT)
Brief Title: Study to Test the Usability of a New Injector to Administer Contrast Media Into Humans for Diagnostic Purposes
Acronym: PERCENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20521
Record Dates: First submitted 2019-02-26; First posted 2019-03-14 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Computed Tomography
Keywords: Contrast-enhanced computed tomography (CECT); Injector

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CT patients_Centargo_1 (Experimental): Adult patients referred for contrast-enhanced computed tomography in study part 1
  Interventions: Device: Centargo injector (BPI 1000045)
- CT-patients_Stellant_1 (Experimental): Adult patients referred for contrast-enhanced computed tomography in study part 1
  Interventions: Device: Stellant MP injector
- CT-patients_Centargo_2 (Experimental): Adult patients referred for contrast-enhanced computed tomography in study part 2 (includes all patients of Arm 1)
  Interventions: Device: Centargo injector (BPI 1000045)

INTERVENTIONS:
Device: Centargo injector (BPI 1000045) — Contrast-enhanced computer tomography conducted with Centargo injector
  Arms: CT patients_Centargo_1; CT-patients_Centargo_2
Device: Stellant MP injector — Contrast-enhanced computer tomography conducted with Stellant MP injector
  Arms: CT-patients_Stellant_1

SUMMARY:
This study investigates if a new medical device, which injects contrast media and flushing solution into humans to increase the visibility of images taken of the human body for diagnostic purposes, is easier to handle, quicker and cheaper than an older injector.

DETAILED DESCRIPTION:
The study compares an investigational injection system (Centargo) for computed tomography (CT) to a currently marketed injection system (Stellant MP) in terms of efficiency, cost, performance and user satisfaction (Part 1). In addition, the reliability of the new injection system Centargo is tested (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects referred for contrast-enhanced computer tomography using a power injector

Exclusion Criteria:

* Pregnant and lactating women
* Subjects with know hypersensitivity to iodinated contrast media
* Subjects with unacceptable renal function per local guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Setup time of CT systems | 1 day
Change time for bottle/ bag containing contrast medium | 1 day
Patient setup time for the multi-patient set per day | 1 day
Teardown time of CT-system | 1 day
Number of multi-patient sets per day | 1 day

SECONDARY OUTCOMES:
Total cost for multi-patients set and disposables per patient and day | 1 day
Reason for change of multi-patient syringe set for the injection of contrast media prior to expiration at 24 hours | 1 day
Volume of unused contrast agent at teardown time | 1 day
Volume of unused saline at teardown time | 1 day
Flow rate of contrast agent through the injector | 1 day
Volume of contrast agent delivered through injector | 1 day
Injector-generated pressure | 1 day
Number of automated system alerts | 1 day
  Incl. alerts due to communication loss, pressure limiting, air detection (Centargo only) and a full waste container (Centrago only).
Radiographer satisfaction with contrast-media injector by study-related questionnaire | Up to 4.5 months
  Questionnaire contains 14 questions on injectors, disposables and software, pertaining to 5 levels of user satisfaction (´Very easy´ to ´Very hard´). Levels of user satisfaction from different questions are not combined.
Number of errors requiring a CT-system reboot | 1 day
  For Centargo only (Part 2)

CONTACTS AND LOCATIONS:
Locations (2):
- Medscan, Merrylands, New South Wales, Australia
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/